CLINICAL TRIAL: NCT02798809
Title: GENOA ORAL GROWTH STUDY: Longitudinal Investigation of Preschool and Primary School Children
Brief Title: GENOA ORAL GROWTH LONGITUDINAL STUDY (GeOrGS)
Acronym: GeOrGS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Genova (Other)
Responsible Party: Principal Investigator, ALESSANDRO UGOLINI, Researcher, University of Genova
Other Study IDs: UGenova
Record Dates: First submitted 2016-06-03; First posted 2016-06-14 (Estimated); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Malocclusion; Dental Caries
MeSH Terms: conditions — Malocclusion; Dental Caries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- GeOrGS cohort: Clinical dental examination of all Children born in 2008 and 2009 in Chivari District (Italy)
  Interventions: Other: Clinical dental examination

INTERVENTIONS:
Other: Clinical dental examination — Clinical dental examination and a questionnaire that was filled out by the parents before each clinical examination.

SUMMARY:
The aim of the study is to follow a group of preschool children from early permanent dentition to determine the prevalence and incidence of caries malocclusions and to investigated the related risk factors as age, gender, ethnic origin and non-nutritive sucking habits, breathing disturbances, allergies, Dietary habits, oral hygiene status and dental care.

DETAILED DESCRIPTION:
Once a year a clinical examination were performed. Data were collected with a questionnaire, that was filled out by the parents before the clinical examination, which included questions on child's clinical history, the type of feeding, the use of baby-bottle, the history of non-nutritive sucking habits (dummy-sucking and digit sucking) and the consent to the clinical examination. Two World Health Organization (WHO) calibrated examiners carried out the clinical examinations. They were blinded to the information collected from the parental questionnaires. Dental examinations were performed in a classroom environment under natural light, using gloves and masks in compliance with the infection control protocol, mouth mirrors and disposable paper rulers to measure overjet and overbite (in millimeters). The occlusion was assessed in centric occlusion and was classified according to Foster and Hamilton criteria [Foster and Hamilton, 1969] Radiographic examination was not performed.

ELIGIBILITY:
Inclusion Criteria:

* children born in 2008 and 2009 in Chiavari District (Italy)

Exclusion Criteria:

* parents' lack of consent
* absence at the date of the visit; no compliance
* orthodontic treatment; marked occlusal wear or early
* loss of primary teeth
* alterations in the number, size and shape of teeth
* syndromes or systemic problems affecting craniofacial growth
* cleft palate.

Ages: 3 Years to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children born in 2008 and 2009 in Chiavari District (Italy)
Sampling Method: Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2012-04-01; Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence (rate %) of Malocclusions and Caries | longitudinal 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Ugolini, DDS, PhD, Principal Investigator — University of Genova
Locations (1):
- Ortohdontic Department - Univesity of Genoa, Genova, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ugolini A, Porro F, Carli F, Agostino P, Silvestrini-Biavati A, Riccomagno E. Probabilistic graphical modelling of early childhood caries development. PLoS One. 2023 Oct 30;18(10):e0293221. doi: 10.1371/journal.pone.0293221. eCollection 2023. PMID 37903153